CLINICAL TRIAL: NCT06529133
Title: The Effect of Dual Task on Postural Control in Children Diagnosed with Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Deniz Tuncer, Assistant professor, Bezmialem Vakif University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024/248
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2024-11

CONDITIONS: Epilepsy; Cognitive Function 1, Social; Balance; Distorted; Children
Keywords: Children; Cognitive dual task; Epilepsy; Postural control
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (Experimental): Healthy children
  Interventions: Other: Evaluation of postural control
- Study Group (Experimental): Children with diagnosed epilepsy
  Interventions: Other: Evaluation of postural control

INTERVENTIONS:
Other: Evaluation of postural control — Postural stability, limits of stability, and modified clinical test of sensory interaction in balance tests will be performed with Biodex Balance System (BBS). 1) Postural Stability: The test will be performed on a stable platform and mean, anterior/posterior and medial/lateral stability indices will be calculated. 2) Limits of Stability: The test will be performed on a static platform and directional control will be evaluated and expressed as a percentage value. 3) Modified Clinical Test of Sensory Interaction in Balance: The test will be performed with a static platform setting on a flat surface with eyes open and eyes closed, on a foam floor with eyes open and eyes closed. Half an hour later, the same tests will be repeated during the cognitive dual task. The cognitive tasks given were counting day-month-season, rhythmic forward and backward counting (counting by 2, 3, 5, 10, etc.), counting words related to a given letter (animal names starting with the letter A, city names, etc.).

SUMMARY:
An individual's postural control is often accompanied by other tasks in daily life, such as cognitive tasks. Cognitive dual task (cognitive dual task) is the ability to perform two or more cognitive and motor activities simultaneously. There are studies in the literature that address the postural control of different patient populations and healthy individuals while performing a cognitive task. To our knowledge, there is no study evaluating the postural control skills of children with epilepsy during a cognitive dual task using dynamic posturography (Biodex). In this respect, it is possible to say that our study constitutes the first study that can contribute to the literature on this subject.

DETAILED DESCRIPTION:
Epilepsy is often characterized by seizures, but may also include additional neurological signs and symptoms that affect the prognosis of the disease. These clinical findings include hypotonia, athetosis, ataxia, inadequate visual-motor functioning, gait abnormalities, balance disorders and learning disabilities. In the literature, it has been reported that individuals with epilepsy who use antiepileptic drugs have more balance problems than those who do not. It is also reported that people with epilepsy exercise less than the general population and have a lower level of functionality compared to their peers. It has also been reported that there is a relationship between age at onset of epilepsy and motor problems.

Executive functions include cognitive processes that support complex, goal-directed behavior, especially in novel situations or situations that require conscious effort. In children diagnosed with epilepsy, visuospatial skills are frequently affected within the scope of executive function.

Postural control mechanism is a complex neural function consisting of the integrated function of sensory input, motor output and modulation by cerebellar and cognitive influences. Lack of coordination and postural instability, motor limitations in patients with epilepsy, and disabilities due to seizures are complaints due to side effects of antiepileptics. Inadequate postural control, which involves the orientation of the body for stabilization in space or task-oriented orientation in harmony with the environment, limits the individual's ability to adapt to the environment or unexpected situations.

An individual's postural control is often accompanied by other tasks in daily life, such as cognitive tasks. Cognitive dual task (cognitive dual task) is the ability to perform two or more cognitive and motor activities simultaneously. There are studies in the literature that address the postural control of different patient populations and healthy individuals while performing a cognitive task. To our knowledge, there is no study evaluating the postural control skills of children with epilepsy during a cognitive dual task using dynamic posturography (Biodex). In this respect, it is possible to say that our study constitutes the first study that can contribute to the literature on this subject.

15 children who are followed up with a diagnosis of epilepsy at Istanbul Faculty of Medicine Child Neurology Polyclinic and who meet the inclusion criteria will be included in the study as the study group, and 15 healthy children in the same age group will be included in the study as the control group. Informed consent will be obtained from each child and parent and the study will be conducted in accordance with the Declaration of Helsinki.

Evaluations and testing of all cases will be carried out in Bezmialem Vakıf University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Pediatric and Cardiac Physiotherapy and Rehabilitation Training and Research Laboratories.

After the demographic information of all children to be included in the study is recorded, they will be informed about the tests to be applied during the cognitive dual task.

Children's postural control abilities will be evaluated with the Biodex Balance System SD (BBS, Biodex Medical Systems, Shirley, NY, USA). With BBS; Postural stability, stability limits and modified sensory integration test (mCTSIB) tests will be performed. Half an hour later, the same tests will be repeated during the cognitive dual task. Cognitive tasks; counting days-months-seasons, rhythmic forward and backward counting (counting by 2s, 3s, 5s, 10s, etc.), counting words related to the specified letter (such as animal names starting with the letter A, city names). Each test will be performed 3 times for 20 seconds.

ELIGIBILITY:
For the study group:

Inclusion Criteria:

1. Being between the ages of 7-16
2. Having been diagnosed with epilepsy
3. Having had a seizure in the last 2 years
4. Being on antiepileptic medication
5. Having a body mass index within normal limits (18.5-24.9 kg/m2)

Exclusion Criteria:

1. Being hypermobile (Beighton score >5 and above)
2. Leg length inequality
3. Having any neurological, rheumatic, musculoskeletal, metabolic and connective tissue disease
4. Pain, deformity or surgical history related to the vertebral column and lower extremity
5. Presence of cognitive, mental and/or serious psychiatric disease
6. Participating in any exercise program or sporting activity in the last six months
7. Hearing and/or vision loss

For the control group:

Inclusion Criteria:

1. Being between the ages of 7-16
2. Having a body mass index within normal limits (18.5-24.9 kg/m2)

Exclusion Criteria:

1. Being hypermobile (Beighton score >5 and above)
2. Leg length inequality
3. Having any neurological, rheumatic, musculoskeletal, metabolic and connective tissue disease
4. Pain, deformity or surgical history related to the vertebral column and lower extremity
5. Presence of cognitive, mental and/or serious psychiatric disease
6. Participating in any exercise program or sporting activity in the last six months
7. Hearing and/or vision loss

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-07-26 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of postural control under two conditions | Day 1
  Postural control abilities of the children will be evaluated with Biodex Balance System (BBS). Half an hour later, the same tests will be repeated during the cognitive dual task.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No